CLINICAL TRIAL: NCT02169297
Title: A Novel Ultrasound-Guided Extrathoracic Sub-Paraspinal Block Utilizing Multi- Perforated Soaker Catheters for Control of Perioperative Pain: A Prospective Randomized Pilot Project in Nuss Patients
Brief Title: Sub-Paraspinal Block in Nuss Patients. A Pilot Project
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 16-10841-002
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-05

CONDITIONS: Pectus Excavatum; Pain, Postoperative
Keywords: Pain Management; Anesthesia: Nerve Block
MeSH Terms: conditions — Funnel Chest; Pain, Postoperative; Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound-Guided Sub-Paraspinal Block (Experimental): Patients allocated to the treatment group received bilateral ultrasound-guided placement of multi-perforated soaker catheter at sub-paraspinal location and an intravenous PCA post-operatively
  Interventions: Procedure: Ultrasound-guided Sub-Paraspinal Block; Procedure: PCA only
- PCA only (Placebo Comparator): Patients allocated to the control group had two sham multi-perforated soaker catheters taped to their back and received intravenous PCA post-operatively
  Interventions: Procedure: PCA only

INTERVENTIONS:
Procedure: Ultrasound-guided Sub-Paraspinal Block — Treatment group received bilateral ultrasound-guided placement of multi-perforated soaker catheter at sub-paraspinal location. Catheter position was considered adequate when live ultrasound imaging confirmed placement directly over the rib surface and lateral to the transverse process at the T2-T10 level. An infusion of ropivacaine 0.2% was started via the On-Q infusion system at a rate of 0.25 mg/kg/hour per catheter (maximum of 8 ml/hr catheter [maximum pump infusion rate]). The local anesthetic infusion was stopped on post-operative day number 3 and the catheters removed.
  Arms: Ultrasound-Guided Sub-Paraspinal Block
Procedure: PCA only — Patients received intravenous PCA post-operatively
  Other Names: Patient-Controlled Analgesia

SUMMARY:
The purpose of this pilot study was to evaluate effectiveness of a novel regional anesthesia technique developed at the investigators institution, as part of a quality improvement initiative, to assist with multilevel thoracic pain control in post-Nuss procedure patients. The investigators hypothesized that the local anesthetic infusion via bilateral multiperforated soaker catheters placed at extrathoracic sub-paraspinal muscle location under ultrasound guidance would significantly improve pain control, as reflected by the decrease in pain intensity score, reduction in opiate requirement and improvement infunctional rehabilitation measure scores in patients who underwent the Nuss procedure for pectus excavatum repair. However, the goal of this pilot study was not to detect a statistically significant difference in the primary outcomes between control and treatment groups (as the number of study subjects was chosen out of necessity of what could be completed within a specified time period), but to estimate the parameters which allows appropriate power and sample size calculations for a future multi-institutional study.

DETAILED DESCRIPTION:
This study underwent initial peer review by the Biomedical Research Committee at Nemours and was awarded internal funding by the Nemours Funding committee. Scientific progress review was conducted annually and was the basis for subsequent year funding.

Ten eligible patients were recruited and allocated into one of two groups according to a computer generated random allocation table: five patients allocated to the treatment group received bilateral ultrasound-guided placement of multi-perforated soaker catheter at sub-paraspinal location and an intravenous PCA post-operatively; five patients allocated to the control group had two sham multi-perforated soaker catheters taped to their back and received intravenous PCA post-operatively. In the treatment group, catheter position was considered adequate when live ultrasound imaging confirmed placement directly over the rib surface and lateral to the transverse process at the T2-T10 level. A 7.5 inch On-Qr multi-perforated catheter was placed via each introducer for patients under 5'7'' (170.18 cm) and a 10" (25.4 cm) catheters was placed for those over 5'7" (170.18 cm). An infusion of ropivacaine 0.2% was started immediately after catheter placement via the On-Q infusion system at a rate of 0.25 mg/kg/hour per catheter (maximum of 8 ml/hr catheter [maximum pump infusion rate]). Maximum total ropivacaine infusion rate was limited to 0.5 mg/kg/hr to avoid toxicity. The local anesthetic infusion was stopped on post-operative day number 3 and the catheters removed.

Catheters were dressed in a way that concealed insertion sites and therefore precluded pain observers from determining group assignment while the pumps appeared to be infusing to blinded viewers. The peri-operative anesthetic and surgical approach were standardized for this study. A single anesthesiologist and surgeon were responsible for the recruitment, anesthesia provision, surgical technique, and multi-perforated soaker catheters insertion. Post-operative pain management was carried out by a group of blinded anesthesiologists according to the post-operative protocol. Three recovery room nurses, six floor nurses and three physical therapists were selected to limit inter observer variability and educated to the post-operative expectations and consistent use of the pain and functional independent measure (FIM) scoring in this patient population. With the exception of the primary investigators, all other personnel were blinded to the patient's group assignment.

The outcomes were evaluated based on the total amount of narcotic per kilogram required, pain scores and functional performance measures derived by physical therapists.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing the Nuss procedure were considered for the study and were approached during their preoperative anesthesia evaluation.

Exclusion Criteria:

* Contraindication to the study medications
* Preexisting chronic pain disorder.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Narcotic Requirement | 48 hours post intervention
  Narcotic requirement was recorded in the PACU and at 6 hour intervals through 48 hours from the time of arrival to PACU

SECONDARY OUTCOMES:
Pain Scores | 48 hours
  Pain scores (FLACC/FACES) were recorded in the PACU and at 6 hour intervals through 48 hours from the time of arrival to PACU

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Bryskin, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Wolfson Children's Hospital, Baptist Medical Center Downtown, Jacksonville, Florida, United States

REFERENCES:
- [Background] Truitt MS, Mooty RC, Amos J, Lorenzo M, Mangram A, Dunn E. Out with the old, in with the new: a novel approach to treating pain associated with rib fractures. World J Surg. 2010 Oct;34(10):2359-62. doi: 10.1007/s00268-010-0651-9. PMID 20567973